CLINICAL TRIAL: NCT00994240
Title: Cure Rates of Superficial Basal Cell Carcinoma Following 1 Versus 3 Cycles of Electrodessication & Curettage: A Randomized Prospective Study
Brief Title: Cure Rates of Superficial Basal Cell Carcinoma (BCC) EDC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment, lack of funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Skin Cancer Foundation (Unknown); Dermatology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2007-0252; PRMC_CO08303 (Other: University of Wisconsin Carbone Cancer Center)
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Superficial Basal Cell Carcinoma
MeSH Terms: interventions — Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ED&C times 3 cycles (Active Comparator)
  Interventions: Procedure: Electrodessication & Curettage
- ED & C times 1 cycle (Active Comparator)
  Interventions: Procedure: Electrodessication & Curettage

INTERVENTIONS:
Procedure: Electrodessication & Curettage — Electrodessication & Curettage 1 or 3 cycles

SUMMARY:
This is a prospective, randomized clinical trial conducted at the Unviersity of Wisconsin (UW) Dermatology Clinic located at 1 S. Park Street, Madison, WI 53715. There are no controls. Subjects meeting eligibility criteria are randomly divided into one of two treatment groups (ED&C x 1 cycle or ED&C x 3 cycles) using computer generated random numbers. One cycle of ED&C is defined according to standard technique currently employed. It involves scraping away the tumor with a curette (ring- shaped instrument) and then burning the curetted site with a small electric needle (electrodessication). During Visit 1, the surgical site is marked, local numbing medication is injected, and 1 or 3 cycles of ED&C is/are performed by board-certified dermatologists or a dermatology resident under the direct supervision of a board certified dermatologist. All follow-up visits (3, 6, 9, and 12 months after Visit 1) include skin evaluations by the physician who performed the ED&C. The lesion site is examined, measured, and photographed for clinical evidence of recurrence, as defined by a new lesion within the previously treated site. If there is evidence of possible tumor recurrence at the treated surgical site during Visit 2, 3, 4 or 5, then the lesion will be biopsied using a shave procedure.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, biopsy proven superficial type basal cell carcinoma (BCC-S) on the trunk and/or extremities
* Age greater than 21
* Women with childbearing potential (including those who are pregnant/lactating)
* Able to provide written informed consent

Exclusion Criteria:

* Aggressive histology on initial biopsy (i.e. morpheaform, infiltrative, desmoplastic, or purely micronodular)
* Prior history of BCC or other skin cancer at the same location
* Lesion > 2 cm
* Patients with basal cell nevus syndrome
* Transplant patients
* Immunocompromised patients
* Recurrent BCC
* Greater than 2 BCC-S on the trunk and/or extremities
* Prisoners
* Allergy to lidocaine or epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Berg, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Department of Dermatology, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ED&C Times 3 Cycles | ED & C Times 1 Cycle
Started | 41 | 44
Completed | 35 | 39
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — study termination | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ED&C Times 3 Cycles | ED & C Times 1 Cycle | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 17 | 24 | 41
Region of Enrollment [Number; unit: participants]
  United States | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: Difference in Cure Rates of Superficial BCC Following One Cycle of ED&C Versus Three Cycles of ED&C.
Description: Clinical evidence of BCC recurrence post treatment
Time Frame: base line, every 3 months until 12 month completion
Population: Study was terminated early due to lack of funding and slow enrollment. Biostatisticians determined insufficient data was available for statistical significance. Primary/lead protocol author is no longer at the institution and no data analysis is intended. Study has been closed with the local IRB and study files archived.
Measure: Number; unit: participants
Arm/Group | ED&C Times 3 Cycles | ED & C Times 1 Cycle
Number analyzed (Participants) | 35 | 39
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | ED&C Times 3 Cycles | ED & C Times 1 Cycle
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 7/41 | 7/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ED&C Times 3 Cycles (N=41) | ED & C Times 1 Cycle (N=44)
itching (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) — mild to moderate itching at the site of treatment
infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — infection at site of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No